CLINICAL TRIAL: NCT02026882
Title: Supreme Laryngeal Mask Use in Urgent Caesarean Section
Brief Title: Supreme LMA Use in Urgent Caesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: QuanZhou Women and Children's Hospital (Other)
Collaborators: KK Women's and Children's Hospital (Other Government)
Responsible Party: Principal Investigator, Wei Yu Yao, Dr, QuanZhou Women and Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-11-11
Record Dates: First submitted 2013-12-31; First posted 2014-01-03 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Airway Morbidity
Keywords: Airway, Caesarean

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Supreme Laryngeal Mask Airway (Other): Supreme Laryngeal Mask Airway with gastric tube. Preoxygenation, rapid sequence induction and cricoid pressure. Induction of general anaesthesia.
  Interventions: Device: Supreme Laryngeal Mask Airway

INTERVENTIONS:
Device: Supreme Laryngeal Mask Airway — Supreme Laryngeal Mask Airway. Preoxygenation, rapid sequence induction and cricoid pressure. Induction of general anaesthesia.

SUMMARY:
The Supreme Laryngeal Mask Airway (SLMA) is a single use supraglottic device that provides a good seal for positive pressure ventilation and good first attempt insertion rate of 98% in low risk patients undergoing elective Caesarean section. It has a double aperture design that facilitates the introduction of an orogastric tube to aspirate gastric contents.

The primary study hypothesis is the first attempt insertion success rate of SLMA use in urgent Caesarean section.

DETAILED DESCRIPTION:
Investigators propose a prospective cohort study to study the first attempt insertion success rate of supreme LMA in general anaesthesia for urgent caesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 50 years old
* American Society of Anesthesiology status 1 or 2
* Weight 40 to 75kg
* Normal airway assessment
* Term pregnancy (36 weeks or more)
* Urgent Caesarean Section

Exclusion Criteria:

* Body mass index (35 or more)
* Difficult airway (Mallampati 4 or abnormal airway assessment)
* Gastrooesophageal reflux

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 584 (Actual)
Dates: Start 2013-12; Primary Completion 2014-12 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
First attempt insertion success rate | 1 hour
  An attempt is defined as insertion and withdrawal of the device from the patient's airway

SECONDARY OUTCOMES:
Time to effective airway placement | 1 hour
  Interval from when the device was picked up until appearance of the first end-tidal carbon dioxide waveform
Aspiration | 1 hour
  Signs of aspiration as evidenced by perioperative hypoxaemia, wheezing or crepitations upon auscultation of lungs or postoperative dyspnoea with chest x ray signs of aspiration
blood on SLMA on removal | 1 hour
  inspection for presence of blood upon removal of SLMA
Sore throat | 1 hour
  Sore throat present in recovery room
Regurgitation | 1 hour
  Gastric contents identified in the mouth with pH less than 4
Seal pressure | 1 hour
  Recorded by closing the adjustable pressure limiting valve and insufflating the closed breathing system with 3L/min fresh gas flow. The peak circuit airway pressure achieved will be recorded.
Gastric aspirate | 1 hour
  Volume of gastric aspirate using gastric tube and pH of gastric aspirate using litmus paper
Neonatal outcomes | 1 hour
  Neonatal birthweight. APGAR score. Umbilical venous cord pH

CONTACTS AND LOCATIONS:
Locations (1):
- Quanzhou Women's and Children's Hospital, Quanzhou, Fujian, China

REFERENCES:
- [Derived] Lim MJ, Tan HS, Tan CW, Li SY, Yao WY, Yuan YJ, Sultana R, Sng BL. The effects of labor on airway outcomes with Supreme laryngeal mask in women undergoing cesarean delivery under general anesthesia: a cohort study. BMC Anesthesiol. 2020 Aug 26;20(1):213. doi: 10.1186/s12871-020-01132-5. PMID 32847548
- [Derived] Tan HS, Li SY, Yao WY, Yuan YJ, Sultana R, Han NR, Sia ATH, Sng BL. Association of Mallampati scoring on airway outcomes in women undergoing general anesthesia with Supreme laryngeal mask airway in cesarean section. BMC Anesthesiol. 2019 Jul 8;19(1):122. doi: 10.1186/s12871-019-0796-5. PMID 31286890
- [Derived] Li SY, Yao WY, Yuan YJ, Tay WS, Han NR, Sultana R, Assam PN, Sia AT, Sng BL. Supreme laryngeal mask airway use in general Anesthesia for category 2 and 3 Cesarean delivery: a prospective cohort study. BMC Anesthesiol. 2017 Dec 19;17(1):169. doi: 10.1186/s12871-017-0460-x. PMID 29258438